CLINICAL TRIAL: NCT01748604
Title: Physical Therapies in the Decongestive Treatment of Lymphedema: A Multicenter, Randomized, Controlled Study.
Brief Title: Physical Therapies in the Decongestive Treatment of Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Forner-Cordero, MD, PhD. (Other)
Responsible Party: Sponsor-Investigator, Isabel Forner-Cordero, MD, PhD., Consultant in Physical Medicine and Rehabilitation at the Lymphedema Unit, Hospital Universitario La Fe
Organization: Hospital Universitario La Fe (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HULaFe-LYMPHEDEMA-04
Record Dates: First submitted 2012-12-06; First posted 2012-12-12 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Primary Lymphedema; Secondary Lymphedema
Keywords: Lymphedema; Physical Therapies; Randomized controlled study; Decongestive lymphatic therapy; Manual lymph drainage; Intermittent pneumatic compression; Multilayer bandages
MeSH Terms: conditions — Lymphedema | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard trimodality therapy with MLD (Active Comparator): Manual Lymphatic Drainage (MLD) followed by intermittent pneumatic compression (IPC) and followed by multilayer, multicomponent bandages (MB) until next day.
  Interventions: Other: Manual Lymphatic Drainage (MLD); Device: Generic intermittent pneumatic compression Device (IPC); Other: multilayer, multicomponent bandages (MB)
- Trimodality therapy with LPD (Experimental): Pneumatic massage with Lymphapress-Plus(TM) device (LPD) followed by intermittent pneumatic compression (IPC) and followed by multilayer, multicomponent bandages (MB) until next day
  Interventions: Device: Generic intermittent pneumatic compression Device (IPC); Other: multilayer, multicomponent bandages (MB); Device: Lymphapress-Plus(TM) device (LPD)
- Bimodality therapy without MLD (Experimental): intermittent pneumatic compression (IPC) followed by multilayer, multicomponent bandages (MB) until next day.
  Interventions: Device: Generic intermittent pneumatic compression Device (IPC); Other: multilayer, multicomponent bandages (MB)

INTERVENTIONS:
Other: Manual Lymphatic Drainage (MLD) — MLD with Földi's technique by an expert therapist during 45 minutes
  Arms: Standard trimodality therapy with MLD
Device: Generic intermittent pneumatic compression Device (IPC) — Generic intermittent pneumatic compression with multicompartmental pump between 50 to 80 mmHg during 30 minutes.
Other: multilayer, multicomponent bandages (MB) — multilayer, multicomponent bandages (MB) until next day.
Device: Lymphapress-Plus(TM) device (LPD) — Pneumatic massage with Lymphapress-Plus(TM)device that was lent during the duration of the study during 20 minutes.
  Arms: Trimodality therapy with LPD

SUMMARY:
The purpose of this multicenter randomised controlled study is to determine whether manual lymphatic drainage (MLD) brings any benefit when added to intermittent pneumatic compression (IPC) plus multilayer, multicomponent bandages (MB) in the decongestive lymphatic therapy (DLT) in patients with lymphedema

DETAILED DESCRIPTION:
Study Design: the study was a multicenter, randomized controlled study conducted at three university hospitals in Spain. Potential subjects were identified at Rehabilitation Department where physicians were responsible for screening subjects for eligibility and enrolling into the study.

Patients that fulfilled the inclusion criteria and signed up the informed consent were stratified within 2 stratums, upper and lower limb lymphedema, and then were randomized to one of the three treatment groups.

The type of randomization was a total randomization with ratio 1:1:1 and the method used to generate the random allocation sequence was a computer-generated random numbers table. Adequate randomization includes calling a central office once eligibility has been determined.

The physicians that assessed the outcome and the statistic who analyzed de data were blinded to the subjects' treatment assignment.

The study was approved by the Research Ethics Committee of the University Hospital La Fe. It was conducted according to the ethical principles laid down in the declaration of Helsinki (52nd World Medical Association General Assembly, Edinburgh, Scotland, October 2000) and the rules of best clinical practice.

Treatment Regimens: Patients were randomized to one of the following treatment groups:

* Group A or control group: Manual Lymphatic Drainage (MLD) with Földi's technique by an expert therapist during 45 minutes; intermittent pneumatic compression (IPC) with multicompartmental pump between 50 to 80 mmHg during 30 minutes, followed by multilayer, multicomponent bandages (MB) until next day.
* Group B: Pneumatic massage with Lymphapress-Plus(TM) device that was lent during the duration of the study during 20 minutes, and was supposed to open the proximal lymphatics at the root of the limb; IPC (50 to 80 mmHg during 30 minutes), followed by MB until next day.
* Group C: IPC (50 to 80 mmHg during 30 minutes) followed by MB until next day.

All patients were planned to receive 20 sessions of treatment (5 per week in consecutive days during 4 consecutive weeks) and were trained in skin care and daily exercises.

After DLT, garments were prescribed and their adaptation was checked to warrant the maintenance of the results. The garments were flat knitted, custom made, generally class 2 (18-21 mmHg) for upper limb, and class 3 (36-46 mmHg) for lower limb.

Sample Size and Statistical analyses: This trial compares the efficacy of two treatment modalities without MLD (experimental group B and C) with a standard trimodal therapy (control group A). The expected effect size in percentage reduction in excess volume (PREV), primary end point, for the control group (MLD+IPC+MB) was defined from the review of literature and was 50 to 70% (mean 60%) with a standard deviation of 20 to 30 (mean 25). Our hypothesis was that there are no differences between experimental and standard treatment.

The required sample size for the study was 177 patients or 59 subjects per group to detect differences greater than or equal 15% in the percentage reduction in excess volume (PREV) between control and experimental groups, if exists; considering differences less than 15% as not clinically significant. It was based on an alpha error of 5% and a power of 90%. We estimated a drop-out rate of 10%. Therefore, 17 patients were added, resulting in a sample size of 194 subjects.

To compare baseline characteristics between three groups we use two-way ANOVA test for continuous variable and Pearson's chi2 for categorical data, to detect potential confounding factors. Outcome data were analyzed utilizing a two-way ANOVA test to assess differences between treatment groups with a 5% level of significance (p≤0.05) and two-tailed tests.

An exploratory subgroup analysis was made to identify factors associated with response (PREV). Factors for initial screening were identified by univariate linear regression model with a p value <0.1. In order to determine the independent predictive factors, a multivariate linear regression analysis was applied.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary lymphedema,
* lymphedema stages II or III
* affecting unilateral upper or lower limb
* Excess volume (EV) > 10%

Exclusion Criteria:

* malignancy or active neoplasm disease or lack of information about it.
* active lymphangitis
* known contraindications for Decongestive Lymphatic Therapy (DLT): renal insufficiency, uncontrolled hypertension, cardiac disease and venous thrombosis.
* a course of DLT during last year.
* anything that could alter the patient's capability to consent truly to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2004-02; Primary Completion 2010-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in Excess Volume (PREV) | at 10 sessions of DLT (2 weeks), at 20 sessions of DLT (4 weeks) and at 1, 6 and 12 months after the end of DLT
  It is obtained with the following formula: [(Initial EV - Final EV)/ Initial EV] x 100; where Excess Volume (EV) is the difference between Lymphedematous (VL) and Healthy limb volume (VH).
  Volumes were calculated with tape perimeter measurements (C) taken from the dorsum of the hand (C1) and repeated for every 4 cm proximally until the axilla (Cn), using Kuhnke formula, as the disk model is considered the method of choice in clinical practice.
  We assessed the change from baseline in PREV during Decongestive Lymphedema Treatment (DLT)and during 12 months of follow-up after DLT.

SECONDARY OUTCOMES:
the Percentage of Volume reduction (PRV) | at 10 sessions of DLT (2 weeks), at 20 sessions of DLT (4 weeks) and at 1, 6 and 12 months after the end of DLT
  it was calculated with the following formula: [(Initial VL - Final VL)/ Initial VL] x 100.
  We assessed the change from baseline in PRV during Decongestive Lymphedema Treatment (DLT)and during 12 months of follow-up after DLT.

OTHER OUTCOMES:
Adverse events related to the treatment | at 10 sessions of DLT (2 weeks), at 20 sessions of DLT (4 weeks) and at 1, 6 and 12 months after the end of DLT
  Discomfort Lymphangitis attacks Edema displacement Fibrosclerotic ring Loss of mobility

CONTACTS AND LOCATIONS:
Overall Officials: Isabel I Forner-Cordero, MD, Phd, Study Director — University Hospital La Fe; Jose J Muñoz-Langa, MD, Phd, Principal Investigator — University Hospital Dr Peset
Locations (1):
- University Hospital La Fe, Valencia, Valencia, Spain

REFERENCES:
- [Background] Johansson K, Lie E, Ekdahl C, Lindfeldt J. A randomized study comparing manual lymph drainage with sequential pneumatic compression for treatment of postoperative arm lymphedema. Lymphology. 1998 Jun;31(2):56-64. PMID 9664269
- [Background] McNeely ML, Magee DJ, Lees AW, Bagnall KM, Haykowsky M, Hanson J. The addition of manual lymph drainage to compression therapy for breast cancer related lymphedema: a randomized controlled trial. Breast Cancer Res Treat. 2004 Jul;86(2):95-106. doi: 10.1023/B:BREA.0000032978.67677.9f. PMID 15319562
- [Background] Badger C, Preston N, Seers K, Mortimer P. Physical therapies for reducing and controlling lymphoedema of the limbs. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003141. doi: 10.1002/14651858.CD003141.pub2. PMID 15495042